CLINICAL TRIAL: NCT01020422
Title: Sexuality and Depression Predictors Among Breast Hypertrophy Women Undergoing Reduction Mammaplasty
Brief Title: Sexuality After Reduction Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Francescato Veiga (Other)
Collaborators: Universidade do Vale do Sapucai (Other)
Responsible Party: Sponsor-Investigator, Daniela Francescato Veiga, Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Dinter 02
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Sexual Function; Depression
Keywords: breast hypertrophy; mammaplasty; sexuality; depression
MeSH Terms: conditions — Depression; Gigantomastia; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast hypertrophy (No Intervention): Patients with macromastia will be evaluated in regard to sexual function and depression predictors at 3 moments: initial interview, after 3 months and after 6 months
- Reduction Mammaplasty (Experimental): Breast hypertrophy patients randomized to this group will immediately be scheduled for reduction mammaplasty and will be will be evaluated in regard to sexual function and depression predictors preoperatively and 3 and 6 months postoperatively
  Interventions: Procedure: Reduction mammaplasty

INTERVENTIONS:
Procedure: Reduction mammaplasty — Sexual function of patients undergoing reduction mammaplasty will be assessed by the Female Sexual Function Index (FSFI) preoperatively and 3 and 6 months postoperatively.
  Other Names: Breast reduction
  Arms: Reduction Mammaplasty

SUMMARY:
The aim of this study is to determine the impact of reduction mammaplasty on sexuality and depression predictors in women with macromastia.

DETAILED DESCRIPTION:
Breast hypertrophy is a common condition among women. Reduction mammaplasty is an effective and well established procedure performed for the relief discomfort associated with breast hypertrophy. Female breasts play an important role in sexuality, thus, the main purpose of this study is to determine whether reduction mammaplasty could influence sexual function and depression predictors on women with breast hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* breast hypertrophy
* candidate to reduction mammaplasty
* healthy volunteer with normal volume breasts (control group)
* body mass index under 30Kg/m2

Exclusion Criteria:

* pregnancy, delivery or breast feeding during the last 12 months
* body mass index over 30Kg/m2
* breast cancer history
* previous breast surgery
* hard smoking

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Sexual function | 6 months
  Sexual function will be assessed by the Female Sexual Function Index (FSFI), pre and 6 months postoperatively.

SECONDARY OUTCOMES:
depression predictors | 6 months
  Depression predictors will me assessed by the Beck Depression Inventory (BDI) pre- and 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia N Beraldo, PhD, Principal Investigator — UNIFESP and UNIVAS; Daniela F Veiga, MD, PhD, Study Director — UNIFESP and UNIVAS; Lydia M Ferreira, MD, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital das Clínicas Samuel Libânio - UNIVÁS, Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Background] Garcia ES, Veiga DF, Sabino-Neto M, Beraldo Cardoso FN, Batista IO, Leme RM, Cabral IV, Novo NF, Ferreira LM. Sensitivity of the Nipple-Areola Complex and Sexual Function Following Reduction Mammaplasty. Aesthet Surg J. 2015 Sep;35(7):NP193-202. doi: 10.1093/asj/sjv034. PMID 26319082
- [Result] Beraldo FN, Veiga DF, Veiga-Filho J, Garcia ES, Vilas-Boas GS, Juliano Y, Sabino-Neto M, Ferreira LM. Sexual Function and Depression Outcomes Among Breast Hypertrophy Patients Undergoing Reduction Mammaplasty: A Randomized Controlled Trial. Ann Plast Surg. 2016 Apr;76(4):379-82. doi: 10.1097/SAP.0000000000000380. PMID 25536204